CLINICAL TRIAL: NCT04071015
Title: Comparison of Continuous Non-Invasive Blood Pressure Measurement Using the Wireless Cuffless Biobeat Monitor with an Invasive Arterial Line Catheter
Brief Title: Comparison of Non-Invasive Blood Pressure (NIBP) Using the Biobeat Device with an Invasive Arterial Line Catheter
Status: Recruiting | Type: Observational
Sponsor: Biobeat Technologies Ltd. (Industry)
Collaborators: The Chaim Sheba Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: Biobeat003
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure; Heart Diseases
Keywords: vital signs; blood pressure; cardiac surgery; non-invasive monitoring
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Non-invasive monitoring — Comparing blood pressure measurement using the Biobeat non-invasive monitor to arterial line.

SUMMARY:
In this clinical study the investigators will compare blood pressure measurements obtained using the non-invasive, wireless Biobeat monitoring device (both a wrist watch and a patch configuration) to an invasive arterial line catheter (radial or femoral) and a Swan Ganz Catheter in 20 patients immediately after cardiac surgery, at the cardiac intensive care unit.

DETAILED DESCRIPTION:
The Biobeat non-invasive, wireless monitoring device is based on reflective photoplethysmograph (PPG) technology. It measures several vital signs, including blood pressure, stroke volume, pulse rate, pulse pressure, heart rate variability, respiratory rate, saturation, cardiac output, cardiac index, and more. The data is transmitted to Biobeat's application (in both Apple and Google Play), and is available on the individual's cellular phone, tablet, or as a full monitoring system in a hospital department. The aim of this study is to compare the Biobeat monitor with the invasive method of blood pressure measurement, an arterial line, and a Swan Ganz catheter for measurements of cardiac output and stroke volume. The study population includes 20 patients undergoing cardiac surgery. As per local protocol, each one of the participants will come out from the operating room with an arterial line, some will also have a Swan Ganz catheter. Once in the intensive care unit, the investigators will attach the Biobeat non-invasive monitor (both a wristwatch and a patch), these two configurations are identical in terms of the monitoring system), and monitor the participants for 4 hours. Though both methods are continuous, the investigators will record the vital signs every 15 minutes during the 4 hours of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above patients of both sexes arriving immediately after cardiac surgery to the intensive care unit with a radial/femoral arterial line and or a Swan Ganz catheter and in need for blood pressure monitoring.

Exclusion Criteria:

* Refusal to participate

  * Patients with no need or no technical capability to have an arterial line
  * Pregnant women
  * Individuals under the age of 18 years
  * Patients with lack of judgment/mental illness
  * Patients working in the Sheba Medical Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients immediately after cardiac surgery arriving to the intensive care unit, and connected to an arterial line and or a Swan Ganz catheter transducer. Usually the arterial line is left for 24 hours. Right after arrival and once connected to an arterial line, the participants will be connected to the Biobeat monitor (both wristwatch or a patch). Vital signs will be monitored for 4 hours, and recorded every 15 minutes, for comparison. After 4 hours, the Biobeat monitor will be disconnected.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Level of accordance between the Biobeat monitor and the arterial line | 4 hours per individual
  Comparing blood pressure measurements of the Biobeat device with those of the arterial line. Both systolic blood pressure and diastolic blood pressure will be assessed during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Kachel, MD, Principal Investigator — The Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel
Locations (1):
- The Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
The investigators would probably share the results showing the level of agreement between the two measurement methods, but it will not be an individual data, rather the whole group, without any personal data included.

REFERENCES:
- [Derived] Hellou E, Jamal T, Zuroff E, Kalhor P, Delgado-Lelievre M, Manzato M, Lerman LO, Lerman A, Kachel E, Zoghby Z. Performance of a cuffless photoplethysmography-based device for continuous monitoring of blood pressure after cardiac surgery: a preliminary validation study. J Hum Hypertens. 2025 Dec;39(12):894-902. doi: 10.1038/s41371-025-01082-w. Epub 2025 Oct 18. PMID 41109863